CLINICAL TRIAL: NCT01796496
Title: Short-term Effect of Manipulative Therapy Techniques in People With Chronic Low Back Pain: A Randomized Controlled Trial.
Brief Title: Manipulative Therapy Techniques to Treat Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Collaborators: Universidad de Granada (Other); Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, Lecturer-PhD, Universidad de Almeria
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: UAL-1
Record Dates: First submitted 2013-02-20; First posted 2013-02-21 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2013-11

CONDITIONS: Low Back Pain; Chronic Disease
Keywords: Low back pain.; Manipulative therapy techniques.; Randomized controlled trial.; Chronic pain.
MeSH Terms: conditions — Low Back Pain; Chronic Disease; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manipulative Therapy Techniques (Experimental): Manipulative Therapy Techniques involve three techniques on lumbar and sacral areas. This protocol will be administered one a week for 3 weeks.
  Interventions: Other: Manipulative Therapy Techniques
- Functional Technique (Active Comparator): Manipulative Therapy Technique involves one technique on lumbar area. This protocol will be administered one a week for 3 weeks.
  Interventions: Other: Functional Technique

INTERVENTIONS:
Other: Manipulative Therapy Techniques — * Global Technical bilateral pelvis: The technique involves inserting a small spine rotation and make a slack in three stages.
  * Indirect technique of lumbar roll in rotation for bilateral L3: to reduce the slack and make the body drop simultaneously, together with a high speed contraction pectoral muscles and triceps, iliac crest leading caudad which produces a rotation of the vertebra underlying joint space opening.
  * Dog-technic on D12: this technique reduces the slack in the abdomen toward the hand in contact with D12. Next, the therapist conducted a thrust in the direction of the reduction.
  Arms: Manipulative Therapy Techniques
Other: Functional Technique — The therapist presses the two anterior superior iliac spines to open the back of the pelvis, this maintained throughout the technique. Then patient is asked to breathe deeply and exhale, sacrum makes a flexion-extension respectively. These movements should be symmetrical and of equal duration in time.
  Arms: Functional Technique

SUMMARY:
The purpose of this study is to analyze the effectiveness of a three manipulative therapy techniques in People with Chronic Low Back Pain.

DETAILED DESCRIPTION:
Objective: To analyze the effectiveness of a three manipulative therapy techniques in individuals with chronic non-specific low back pain of mechanical etiology.

Design: Randomized clinical trial. Setting: Almeria, South Spain. Participants: Sixty two with chronic non-specific low back pain will be randomly assigned to an experimental or control group.

Intervention: For 3-week, the experimental group will undergo treatment comprising 3 sessions (1/week) of manipulative therapy techniques in the lumbar and sacral areas, and the control group will receive a functional technique in the lumbar area.

Main Outcome Measures: Oswestry disability index, pain visual analogue scale, Tampa scale for kinesiophobia, Roland-Morris disability questionnaire, McQuade test, quality of life scores and the range of trunk anteflexion motion, which were all assessed before the treatment and immediately after the last treatment session.

The primary outcome measure is the change in the RMDQ score at the end of the 3 weeks study period. A difference of 2.5 point is considered to be the minimum clinically important difference in the RMDQ score. A sample size of 62 patients (31 per group) would enable detection of a 2.5 point difference between groups given 80-90% power, a 5% (two-tailed) significance level, and a conservative standard derivation of 5 points. Key baseline demographic variables and clinical measure scores will be compared between groups by using independent Student t tests for continuous data and chi-square tests for categorical data. Separate 2x2 mixed model ANOVA with repeated measurements for the time factor need to be conducted in order to test between-groups differences in visual analogue scale, McQuade test, range of trunk anteflexion motion, Oswestry disability index, Roland Morris disability questionnaire, Tampa scale for kinesiophobia, and quality of life as the dependent variables, with group (functional technique or three manipulative therapy techniques) as the between subjects variable and time (baseline, post-treatment). A paired t-test will perform to test within-group differences in score changes from pre- to post-treatment. Effect size will test using Cohen's d. p = 0.05 will be considered significant in all tests.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain for ≥ 3 months.
* Score ≥4 on the Roland Morris disability questionnaire.
* No undergoing another physical therapy treatment.
* Inability to achieve lumbar muscle flexion-relaxation in trunk flexion

Exclusion Criteria:

* Clinical signs of radiculopathy.
* Presence of lumbar stenosis.
* Fibromyalgia.
* Spondylolisthesis.
* History of spinal surgery.
* Treatment with corticosteroids in the past two weeks.
* Disease of the central or peripheral nervous system.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Roland Morris Disability Questionnaire (RMDQ) | At baseline, 3 weeks and 7 weeks
  The Roland Morris disability questionnaire is a self-administered disability measurement scored on a 24-point scale from 0 = no disability to 24 = severe disability.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | At baseline, 3 weeks and 7 weeks
  The Oswestry disability index evaluates daily life activity limitations in 10 dimensions, each scored on a 6-point scale (0-5 points); the total points scored are expressed as a percentage, used to classify individuals as minimally disabled (0-10%), moderately disabled (20-40%), severely disabled (40-60%), crippled (60-80%), or bedbound (80-100%).
Visual Analogue Scale (VAS) | At baseline, 3 weeks and 7 weeks
  The visual analogue scale for pain intensity ranged from 0 = no pain to 10 = worst imaginable pain.
Tampa Scale for Kinesiophobia (TSK) | At baseline, 3 weeks and 7 weeks
  The Tampa Scale for Kinesiophobia comprises 17 items on the fear of movement or recurrent lesion, each scored on a 4-point Likert scale from "completely disagree" to "completely agree".
Quality of Life | At baseline, 3 weeks and 7 weeks
  SF-36 Health Questionnaire scores range from 0 to 100% and indicate the self-perceived health-related quality of life.
Isometric Resistance of Abdominal Muscles | At baseline, 3 weeks and 7 weeks
  The McQuade test measures the isometric resistance of abdominal muscles in seconds.
Lumbar Mobility in Flexion | At baseline, 3 weeks and 7 weeks
  Lumbar mobility in flexion was determined by measuring the distance from the tip of the third finger to the floor with a tape measure.

CONTACTS AND LOCATIONS:
Overall Officials: Adelaida M Castro-Sánchez, PhD, Study Director — Universidad de Almeria
Locations (1):
- Adelaida María Castro-Sánchez, Almería, Almeria, Spain

REFERENCES:
- [Background] Schafer A, Gartner-Tschacher N, Schottker-Koniger T. [Subgroup-specific therapy of low back pain: description and validity of two classification systems]. Orthopade. 2013 Feb;42(2):90-9. doi: 10.1007/s00132-012-2041-5. German. PMID 23370728
- [Background] Rodeghero JR, Denninger TR, Ross MD. Abdominal pain in physical therapy practice: 3 patient cases. J Orthop Sports Phys Ther. 2013 Feb;43(2):44-53. doi: 10.2519/jospt.2013.4408. Epub 2013 Jan 14. PMID 23322025
- [Background] Muir JM. Partial lumbosacral transitional vertebrae: 2 cases of unilateral sacralization. J Chiropr Med. 2012 Jun;11(2):77-83. doi: 10.1016/j.jcm.2011.12.002. PMID 23204950
- [Background] Shum GL, Tsung BY, Lee RY. The immediate effect of posteroanterior mobilization on reducing back pain and the stiffness of the lumbar spine. Arch Phys Med Rehabil. 2013 Apr;94(4):673-9. doi: 10.1016/j.apmr.2012.11.020. Epub 2012 Nov 23. PMID 23178541
- [Background] Falco FJ, Manchikanti L, Datta S, Sehgal N, Geffert S, Onyewu O, Zhu J, Coubarous S, Hameed M, Ward SP, Sharma M, Hameed H, Singh V, Boswell MV. An update of the effectiveness of therapeutic lumbar facet joint interventions. Pain Physician. 2012 Nov-Dec;15(6):E909-53. PMID 23159980
- [Background] Williams JM, Haq I, Lee RY. The effect of pain relief on dynamic changes in lumbar curvature. Man Ther. 2013 Apr;18(2):149-54. doi: 10.1016/j.math.2012.09.004. Epub 2012 Oct 9. PMID 23058448
- [Background] Williams JM, Haq I, Lee RY. A novel approach to the clinical evaluation of differential kinematics of the lumbar spine. Man Ther. 2013 Apr;18(2):130-5. doi: 10.1016/j.math.2012.08.003. Epub 2012 Oct 6. PMID 23047044
- [Background] Hendrick P, Mani R, Bishop A, Milosavljevic S, Schneiders AG. Therapist knowledge, adherence and use of low back pain guidelines to inform clinical decisions--a national survey of manipulative and sports physiotherapists in New Zealand. Man Ther. 2013 Apr;18(2):136-42. doi: 10.1016/j.math.2012.09.002. Epub 2012 Oct 6. PMID 23047043
- [Background] Cook C, Learman K, Showalter C, Kabbaz V, O'Halloran B. Early use of thrust manipulation versus non-thrust manipulation: a randomized clinical trial. Man Ther. 2013 Jun;18(3):191-8. doi: 10.1016/j.math.2012.08.005. Epub 2012 Oct 2. PMID 23040656
- [Background] Carlsson H, Rasmussen-Barr E. Clinical screening tests for assessing movement control in non-specific low-back pain. A systematic review of intra- and inter-observer reliability studies. Man Ther. 2013 Apr;18(2):103-10. doi: 10.1016/j.math.2012.08.004. Epub 2012 Sep 25. PMID 23018080
- [Background] Rubinstein SM, Terwee CB, Assendelft WJ, de Boer MR, van Tulder MW. Spinal manipulative therapy for acute low-back pain. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD008880. doi: 10.1002/14651858.CD008880.pub2. PMID 22972127
- [Background] Marlowe D. Complementary and alternative medicine treatments for low back pain. Prim Care. 2012 Sep;39(3):533-46. doi: 10.1016/j.pop.2012.06.008. Epub 2012 Jul 30. PMID 22958563
- [Background] Guild DG. Mechanical therapy for low back pain. Prim Care. 2012 Sep;39(3):511-6. doi: 10.1016/j.pop.2012.06.006. PMID 22958560
- [Background] Balthazard P, de Goumoens P, Rivier G, Demeulenaere P, Ballabeni P, Deriaz O. Manual therapy followed by specific active exercises versus a placebo followed by specific active exercises on the improvement of functional disability in patients with chronic non specific low back pain: a randomized controlled trial. BMC Musculoskelet Disord. 2012 Aug 28;13:162. doi: 10.1186/1471-2474-13-162. PMID 22925609
- [Background] Tufo A, Desai GJ, Cox WJ. Psoas syndrome: a frequently missed diagnosis. J Am Osteopath Assoc. 2012 Aug;112(8):522-8. doi: 10.7556/jaoa.2012.112.8.522. PMID 22904251
- [Background] Peterson CK, Bolton J, Humphreys BK. Predictors of improvement in patients with acute and chronic low back pain undergoing chiropractic treatment. J Manipulative Physiol Ther. 2012 Sep;35(7):525-33. doi: 10.1016/j.jmpt.2012.06.003. Epub 2012 Jul 31. PMID 22858233
- [Background] Licciardone JC, Kearns CM. Somatic dysfunction and its association with chronic low back pain, back-specific functioning, and general health: results from the OSTEOPATHIC Trial. J Am Osteopath Assoc. 2012 Jul;112(7):420-8. PMID 22802542
- [Background] Mazaheri M, Coenen P, Parnianpour M, Kiers H, van Dieen JH. Low back pain and postural sway during quiet standing with and without sensory manipulation: a systematic review. Gait Posture. 2013 Jan;37(1):12-22. doi: 10.1016/j.gaitpost.2012.06.013. Epub 2012 Jul 15. PMID 22796243
- [Background] Alpert BS. Exercise in sickle cell anemia. Pediatr Cardiol. 1990 Oct;11(4):227. doi: 10.1007/BF02238375. No abstract available. PMID 2274454
- [Background] Vora RN, Barron BA, Almudevar A, Utell MJ. Work-related chronic low back pain-return-to-work outcomes after referral to interventional pain and spine clinics. Spine (Phila Pa 1976). 2012 Sep 15;37(20):E1282-9. doi: 10.1097/BRS.0b013e318265a930. PMID 22739674
- [Background] Tozzi P, Bongiorno D, Vitturini C. Low back pain and kidney mobility: local osteopathic fascial manipulation decreases pain perception and improves renal mobility. J Bodyw Mov Ther. 2012 Jul;16(3):381-391. doi: 10.1016/j.jbmt.2012.02.001. Epub 2012 Mar 3. PMID 22703751
- [Background] Vismara L, Cimolin V, Menegoni F, Zaina F, Galli M, Negrini S, Villa V, Capodaglio P. Osteopathic manipulative treatment in obese patients with chronic low back pain: a pilot study. Man Ther. 2012 Oct;17(5):451-5. doi: 10.1016/j.math.2012.05.002. Epub 2012 May 31. PMID 22658268
- [Background] Hansen H, Manchikanti L, Simopoulos TT, Christo PJ, Gupta S, Smith HS, Hameed H, Cohen SP. A systematic evaluation of the therapeutic effectiveness of sacroiliac joint interventions. Pain Physician. 2012 May-Jun;15(3):E247-78. PMID 22622913
- [Background] Day JM, Nitz AJ. The effect of muscle energy techniques on disability and pain scores in individuals with low back pain. J Sport Rehabil. 2012 May;21(2):194-8. doi: 10.1123/jsr.21.2.194. PMID 22622384
- [Background] Cohen BL. Emerging technologies in the field of healthcare: enhancing the interface to the medical professional. Ann Acad Med Singap. 1990 Sep;19(5):627-39. PMID 2260817
- [Background] Parker J, Heinking KP, Kappler RE. Efficacy of osteopathic manipulative treatment for low back pain in euhydrated and hypohydrated conditions: a randomized crossover trial. J Am Osteopath Assoc. 2012 May;112(5):276-84. PMID 22582197